CLINICAL TRIAL: NCT07317674
Title: The Effect of Nipple Stimulation Combined With Foley Balloon Catheter on Bishop Score and Induction-to-delivery Interval: a Prospective Randomized Trial
Brief Title: Combined Nipple Stimulation and Foley Balloon for Cervical Ripening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr Raneen Abu Shqara, Head of MFMU, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHR-0186-25
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Induction of Labor; Cervical Ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley Balloon Catheter Combined With Nipple Stimulation (Experimental): Participants in this arm will undergo cervical ripening using a single-balloon Foley catheter. One hour after catheter insertion, nipple stimulation will be initiated using a breast pump according to a standardized protocol (15 minutes per breast, alternating with 15-minute rest periods, for up to 6 hours or until active labor, membrane rupture, uterine tachysystole, or non-reassuring fetal heart rate occurs).
  Interventions: Procedure: Foley balloon catheter with nipple stimulation
- Foley Balloon Catheter Alone (Active Comparator): Participants in this arm will undergo cervical ripening using a single-balloon Foley catheter alone, without nipple stimulation. Labor management following catheter insertion and removal will follow standard institutional protocols.
  Interventions: Procedure: Mechanical cervical ripening with Foley catheter

INTERVENTIONS:
Procedure: Foley balloon catheter with nipple stimulation — Mechanical cervical ripening will be performed using a single-balloon Foley catheter inserted transcervically under sterile conditions. The catheter balloon will be positioned above the internal cervical os and inflated with 60 mL of sterile saline solution. The catheter will remain in place for up to 12 hours or until spontaneous expulsion, onset of active labor, rupture of membranes, uterine tachysystole, or non-reassuring fetal heart rate tracing, whichever occurs first.
  In participants randomized to the intervention arm, cervical ripening with the Foley catheter will be combined with nipple stimulation using an electric breast pump according to a standardized protocol, beginning one hour after catheter insertion. Participants in the control arm will undergo cervical ripening with the Foley catheter alone, without nipple stimulation.
  Cervical status will be assessed before catheter insertion and after catheter removal using the Bishop score. Subsequent labor management will follow
  Arms: Foley Balloon Catheter Combined With Nipple Stimulation
Procedure: Mechanical cervical ripening with Foley catheter — Mechanical cervical ripening will be performed using a single-balloon Foley catheter inserted transcervically under sterile conditions. The catheter balloon will be positioned above the internal cervical os and inflated with 60 mL of sterile saline solution. The catheter will remain in place for up to 12 hours or until spontaneous expulsion, onset of active labor, rupture of membranes, uterine tachysystole, or non-reassuring fetal heart rate tracing, whichever occurs first.
  Arms: Foley Balloon Catheter Alone

SUMMARY:
Labor induction rates have increased substantially worldwide, and successful cervical ripening remains a key determinant of induction outcomes. Mechanical cervical ripening with a Foley balloon catheter is widely used and considered safe, while nipple stimulation promotes endogenous oxytocin release and represents a physiologic method for stimulating uterine contractions. However, the combined effect of nipple stimulation and balloon catheter use has not been systematically evaluated.

This prospective, randomized, double-blinded controlled trial will assess whether the addition of nipple stimulation to Foley balloon catheter cervical ripening improves Bishop score and shortens the induction-to-delivery interval compared with balloon catheter alone. Term pregnant patients (37-42 weeks' gestation) with a singleton, cephalic pregnancy and an unfavorable cervix (Bishop score <6) requiring labor induction will be randomized to receive either Foley balloon catheter plus standardized nipple stimulation or Foley balloon catheter alone.

The primary outcomes are change in Bishop score after catheter removal and time from catheter insertion to delivery. Secondary outcomes include need for additional induction methods, mode of delivery, maternal and neonatal outcomes, pain, patient satisfaction, and breastfeeding rates. The study aims to evaluate the efficacy and safety of incorporating a physiologic intervention into standard mechanical cervical ripening.

DETAILED DESCRIPTION:
Rates of labor induction have increased substantially in recent decades in Israel and worldwide. Cervical ripening is a critical component of successful labor induction, and an unfavorable cervix, as reflected by a low Bishop score, is associated with prolonged induction, increased need for additional interventions, and higher rates of operative delivery. Mechanical methods, particularly the Foley balloon catheter, are commonly used for cervical ripening due to their effectiveness and favorable safety profile, including a lower risk of uterine tachysystole compared with pharmacologic agents.

Nipple stimulation is a non-pharmacologic, physiologic method that promotes endogenous oxytocin release and uterine contractions, mimicking spontaneous labor. Prior studies have suggested that nipple stimulation may reduce the need for exogenous oxytocin and lower the incidence of uterine hyperstimulation, while achieving comparable maternal and neonatal outcomes. However, the combined use of nipple stimulation with mechanical cervical ripening has not been systematically evaluated.

This study is a prospective, randomized, double-blinded controlled trial designed to evaluate whether the addition of nipple stimulation to Foley balloon catheter cervical ripening improves cervical readiness and shortens the induction-to-delivery interval compared with Foley balloon catheter alone. Eligible participants are term pregnant patients (37-42 weeks' gestation) with singleton, cephalic pregnancies, intact membranes, and an unfavorable cervix (Bishop score <6) who require labor induction for standard obstetric indications.

Participants will be randomized in a 1:1 ratio to one of two study groups. The intervention group will undergo cervical ripening with a Foley balloon catheter in combination with a standardized nipple stimulation protocol using a breast pump. Nipple stimulation will begin one hour after catheter insertion and will consist of alternating stimulation of each breast for 15 minutes with 15-minute rest intervals, for up to six hours, at the maximum tolerable intensity. The control group will receive cervical ripening with a Foley balloon catheter alone, with standard obstetric management.

Fetal heart rate monitoring will be performed at regular intervals according to institutional protocols, with increased monitoring as clinically indicated. The balloon catheter will be removed after 12 hours, earlier if spontaneous labor ensues, membranes rupture, uterine tachysystole occurs, or non-reassuring fetal status is suspected.

Primary outcomes include the change in Bishop score following catheter removal and the induction-to-delivery interval. Secondary outcomes include the need for additional induction methods (e.g., oxytocin or prostaglandins), time to active labor, mode of delivery, maternal complications (including intrapartum fever, chorioamnionitis, postpartum hemorrhage, and uterine tachysystole), neonatal outcomes (Apgar scores, umbilical cord pH, NICU admission), maternal pain and satisfaction scores, and breastfeeding rates.

The findings of this study will provide evidence regarding the efficacy and safety of integrating a physiologic intervention with mechanical cervical ripening and may inform future strategies to optimize labor induction while minimizing pharmacologic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals aged ≥18 years
* Singleton pregnancy
* Term gestation (37-42 weeks)
* Cephalic fetal presentation
* Intact membranes
* Bishop score <6 at enrollment
* Medical indication for labor induction

Exclusion Criteria:

* Multiple gestation
* Previous cesarean delivery or uterine surgery
* Contraindication to vaginal delivery
* Major fetal anomalies
* Active labor at enrollment
* Unstable fetal lie or presentation
* Contraindication to Foley balloon catheter insertion
* Conditions precluding nipple stimulation (e.g., local breast infection, prior breast surgery involving the nipple)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to individuals who self-identify as female and are pregnant.
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Induction-to-delivery interval | From Foley balloon catheter insertion until delivery (up to 48 hours)
  Defined as the time (in hours) from Foley balloon catheter insertion until delivery.
Change in Bishop score | From Foley balloon catheter insertion until catheter removal (up to 12 hours)
  Defined as the difference between the Bishop score before Foley balloon catheter insertion and after catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Frank Wolf, Prof., Study Chair — Galilee Medical Center

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. De-identified aggregate data may be presented in scientific publications and presentations in accordance with institutional policies and ethical approvals.

REFERENCES:
- [Result] Kavanagh J, Kelly AJ, Thomas J. Breast stimulation for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003392. doi: 10.1002/14651858.CD003392.pub2. PMID 16034897
- [Result] Abu Shqara R, Goldinfeld G, Assulyn T, Sgayer I, Ganem N, Lowenstein L, Frank Wolf M. Breast stimulation vs low dose oxytocin for labor augmentation in women with a previous cesarean delivery, a randomized controlled trial. Am J Obstet Gynecol MFM. 2025 May;7(5):101658. doi: 10.1016/j.ajogmf.2025.101658. Epub 2025 Mar 5. PMID 40054666
- [Result] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2019 Oct 18;10(10):CD001233. doi: 10.1002/14651858.CD001233.pub3. PMID 31623014